CLINICAL TRIAL: NCT04330235
Title: Evaluating a Healthy Restaurant Kids Meals Policy
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); University of Pennsylvania (Other); Harvard Pilgrim Health Care (Other); University of Minnesota (Other); RTI International (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: HDB-NYC; 1R01HD100983-01 (NIH)
Record Dates: First submitted 2020-01-16; First posted 2020-04-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Children 2-10 years of age dining at fast-food restaurants in New York City and Philadelphia, where a healthy default beverage policy will be enacted.
  Interventions: Other: Healthy Default Kids' Beverage Policy
- Control Group: Children 2-10 years of age dining at fast-food restaurants in northern New Jersey, where a healthy default beverage policy will not be enacted.

INTERVENTIONS:
Other: Healthy Default Kids' Beverage Policy — The healthy default kids' beverage policy requires that all restaurants serve only healthy beverages (water, milk, or 100% juice) instead of sugary beverages as the default beverage with children's meals. The policy has been enacted in New York City and Philadelphia and will go into effect in April 2020.
  Other Names: Healthy Restaurant Kids' Meals Policy; Healthy Default Beverage Policy; Healthy Default Beverage Law; Healthy-by-Default Policy
  Groups: Intervention Group

SUMMARY:
More than a dozen municipalities have passed healthy default kids' beverage policies. These policies seek to reduce child consumption of sugar-sweetened beverages (SSBs) by requiring that restaurants serve only healthy beverages (e.g., water, milk, or 100% juice) instead of SSBs as the default choice with children's meals in restaurants. These policies have potential to meaningfully reduce child SSB consumption. However, there are significant gaps in our knowledge of the effects of healthy default beverage policies on children's health. This study uses a natural experiment to evaluate the effects of a healthy default beverage policy in two U.S. cities, New York City and Philadelphia, on children's fast-food restaurant meal orders and dietary intake. The primary hypothesis is that the policy will reduce children's SSB purchases and consumption, reduce children's total caloric intake, and improve diet quality at the fast-food restaurant meal and on the day of the restaurant meal.

DETAILED DESCRIPTION:
This study uses a quasi-experimental approach to evaluate the effects of a healthy default kids' beverage policy on children's fast-food restaurant meal purchases and dietary intake. Annotated receipt and survey data will be collected from parents purchasing a food or beverage for a child 2-10 years of age at fast-food restaurants. Eligible participants will be asked to participate in a telephone dietary recall the following day. Data will be collected from a repeated cross-section of children in two intervention cities implementing a healthy default kids' beverage policy (New York City and Philadelphia) and a control area not implementing the policy (northern New Jersey) before the policy is implemented and after the policy goes into effect. A difference-in-differences analytic approach will be used to compare the change in children's fast-food restaurant meal orders and dietary intake pre- to post-implementation in the intervention versus control groups. A Holm-Bonferroni correction for multiple comparisons will be applied to p-values for secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older
* Parent or legal guardian of a child 2-10 years of age
* Purchasing at least one food or beverage item for the child at the restaurant (if purchasing foods or beverages for multiple children, only items purchased for the youngest child 2-10 years of age will be included)
* Able to speak and understand English or Spanish

Additional criteria for dietary recalls:

* Parent or legal guardian 18 years of age or older is present for the recall
* If child for whom the restaurant meal was purchased is 6 years of age or older, child is present for the recall
* If child for whom the restaurant meal was purchased is 9 years of age or older, the child is present for the recall and is able to speak and understand English or Spanish

Exclusion Criteria:

* Younger than 18 years of age
* Is not a parent or legal guardian to a child 2-10 years of age
* Is not purchasing one or more food or beverage items for the child at the restaurant
* Does not speak or understand English or Spanish

Additional criteria for dietary recalls:

* Parent or legal guardian is not present for the recall
* The restaurant meal was purchased for a child 6 years of age or older, who is not present for the recall
* Child 9 years of age or older, for whom the restaurant meal was purchased, is not able to speak or understand English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents/legal guardians of children 2-10 years of age will be recruited from fast-food restaurants in Philadelphia, northern New Jersey, and New York City that operate more than one location in both the intervention and control areas, serve kids' meals, and are not compliant with the healthy default kids' beverage policy at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 3480 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline total caloric intake at 24 months | 24 months
  Total calories consumed by the child on the day of the restaurant meal

SECONDARY OUTCOMES:
Change from baseline calories consumed from sugar-sweetened beverages at 24 months | 24 months
  Calories consumed by the child from sugar-sweetened beverages on the day of the restaurant meal
Change from baseline calories consumed from healthy beverages at 24 months | 24 months
  Calories consumed by the child from healthy beverages as defined by NYC/Philadelphia law on the day of the restaurant meal
Change from baseline calories consumed from other unhealthy beverages at 24 months | 24 months
  Calories consumed by the child from unhealthy beverages as defined by NYC/Philadelphia law, excluding sugar-sweetened beverages, on the day of the restaurant meal
Change from baseline Healthy Eating Index 2015 score at 24 months | 24 months
  Child's diet quality, measured using the Healthy Eating Index 2015, on the day of the restaurant meal. The Healthy Eating Index 2015 measures how well a diet aligns with the Dietary Guidelines for Americans. It is measured on a scale from 0-100, where higher scores indicate a healthier diet.
Change from baseline total caloric intake during the restaurant meal at 24 months | 24 months
  Total calories consumed by the child during the restaurant eating occasion
Change from baseline calories consumed from sugar-sweetened beverages during the restaurant meal at 24 months | 24 months
  Calories consumed by the child from sugar-sweetened beverages during the restaurant eating occasion
Change from baseline calories consumed from healthy beverages during the restaurant meal at 24 months | 24 months
  Calories consumed by the child from healthy beverages as defined by NYC/Philadelphia law during the restaurant eating occasion
Change from baseline calories consumed from other unhealthy beverages during the restaurant meal at 24 months | 24 months
  Calories consumed by the child from unhealthy beverages as defined by NYC/Philadelphia law, excluding sugar-sweetened beverages, during the restaurant eating occasion
Change from baseline Healthy Eating Index 2015 score during the restaurant meal at 24 months | 24 months
  Child's diet quality, measured using the Healthy Eating Index 2015, during the restaurant eating occasion. The Healthy Eating Index 2015 measures how well a diet aligns with the Dietary Guidelines for Americans. It is measured on a scale from 0-100, where higher scores indicate a healthier diet.
Change from baseline fluid ounces of sugar-sweetened beverages purchased at 24 months | 24 months
  Fluid ounces of sugar-sweetened beverages purchased for the child at the restaurant
Change from baseline fluid ounces of healthy beverages purchased at 24 months | 24 months
  Fluid ounces of healthy beverages as defined by NYC/Philadelphia law purchased for the child at the restaurant
Change from baseline fluid ounces of other unhealthy beverages purchased at 24 months | 24 months
  Fluid ounces of unhealthy beverages as defined by NYC/Philadelphia law, excluding sugar-sweetened beverages, purchased for the child at the restaurant
Change from baseline frequency of dining at fast food restaurants at 24 months | 24 months
  Number of lunch or dinner meals from fast food restaurants for the child in the past week

OTHER OUTCOMES:
Change from baseline fluid ounces consumed from sugar-sweetened beverages at 24 months | 24 months
  Fluid ounces consumed by the child from sugar-sweetened beverages on the day of the restaurant meal
Change from baseline fluid ounces consumed from healthy beverages at 24 months | 24 months
  Fluid ounces consumed by the child from healthy beverages as defined by NYC/Philadelphia law on the day of the restaurant meal
Change from baseline fluid ounces consumed from other unhealthy beverages at 24 months | 24 months
  Fluid ounces consumed by the child from unhealthy beverages as defined by NYC/Philadelphia law, excluding sugar-sweetened beverages, on the day of the restaurant meal

CONTACTS AND LOCATIONS:
Overall Officials: Alyssa Moran, ScD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Angie Cradock, ScD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- United States (3):
  - University of Minnesota, Minneapolis, Minnesota
  - RTI, International, Research Triangle Park, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided